CLINICAL TRIAL: NCT03734042
Title: Intrauterine Infusion of Platelet-rich Plasma Infusion Before Thawed Embryo Transfer in Repeated Implantation Failure: A Randomized Controlled Study
Brief Title: PRP Intrauterine Infusion in Thawed Embryo Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRPF
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Evaluations
Keywords: Platelet rich plasma; Intrauterine infusion; Thawed embryos; IVF/ICSI cycles
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 2 groups parallel
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP group (Experimental): These patients will receive platelet rich plasma intrauterine infusion at day 11
  Interventions: Biological: Platelet rich plasma intrauterine infusion
- Control group (Placebo Comparator): These patients will receive intrauterine normal saline infusion at day 11
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Platelet rich plasma intrauterine infusion — platelet rich plasma will be prepared, activated then infused by Intrauterine insemination catheter intrauterine at day 11
  Arms: PRP group
Biological: Normal saline — Intrauterine infusion of normal saline at day 11
  Arms: Control group

SUMMARY:
All patients prepared to thawed embryo transfer were classified into 2 groups one group will receive platelet rich plasma (PRP) infusion intrauterine and the other group will not receive platelet rich plasma (PRP) infusion

DETAILED DESCRIPTION:
Patients candidates for Thawed embryo transfer with Repeated implantation failure were recruited from 3 centers and classified into 2 groups:

Group I: Will receive platelet rich plasma (PRP) intrauterine infusion at day 11

Group II: Not receiving platelet rich plasma (PRP)

ELIGIBILITY:
Inclusion Criteria:

* Patients age 20-35 years
* Patients with previous implantation failure
* Patients with thin endometrium<7 mm

Exclusion Criteria:

* Patients older than 40 years
* Patients with fresh embryo transfer
* Patients with abnormal uterine cavity septate, or bicornuate uterus
* Patients with abnormal male factor or tubal factor
* Patients with abnormal embryos grade B or C.
* Patients with immunological disorders as thyroidits or systemic lupus or rheumatoid arthritis

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness | 8 days
  The increase in endometrial thickness at day of ET
Pregnancy rate | 15 days
  Number of cases who got pregnant

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
not allowed